CLINICAL TRIAL: NCT06507046
Title: Robotic Assisted Surgery Comparing Personalized Alignment Versus Mechanical Alignment of Total Knee Arthroplasty - A Randomized Controlled Trial
Brief Title: The personalKNEE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Oslo University Hospital (Other); National Taiwan Normal University (Other); University of Oslo (Other); Sectra AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 738578
Record Dates: First submitted 2024-07-08; First posted 2024-07-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient, nurses and physiotherapists are blinded. Surgeon is of course not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical alignment (Active Comparator): Patients are operated with ROSA robot and mechanical alignment
  Interventions: Procedure: Total knee replacement
- Personalized alignment (Experimental): Patients are operated with ROSA robot and kinematic alignment
  Interventions: Procedure: Total knee replacement

INTERVENTIONS:
Procedure: Total knee replacement — Mechanical or Personalized alignment

SUMMARY:
Robotic knee surgery makes it possible to adopt different alignment philosophies in total knee arthroplasty. The classical operation where the knee is placed in a neutral manner, the so called mechanical alignment, has been used for decades. The kinematical alignment has recently won popularity. With this technique the focus is to render the natural knee anatomy even if this means to end up with a varus or valgus position. In this study, the investigators will compare the mechanical alignment and kinematical alignment and test the patients clinically and with a special CT scan to see if this technique gives equal or better longevity of the implants.

DETAILED DESCRIPTION:
Mechanical alignment (MA) has for many years been the most used surgical alignment technique in total knee arthroplasty (TKA). This means that regardless of constitutional native anatomy (i.e. valgus or varus), one strives to achieve a neutral coronal knee axis on postoperative x-rays (Hip-Knee-Ankle angle, HKA). To achieve MA, the cuts are made perpendicular to the mechanical axis, and subsequent soft tissue balancing is performed if necessary. However, many patients do not have a neutral knee alignment before they develop osteoarthritis. Several authors therefore advocate the personalized alignment (kinematic, KA or functional alignment, FA), where the aim is to restore the patient's original pre-arthritis anatomy and joint line. This means that tibial component placement in varus or valgus is accepted, despite the possible result of a postoperative non-neutral HKA axis. Studies indicate that good clinical results can be achieved in terms of range of motion (ROM) and patient reported outcome measures (PROMs) with these techniques, but it has not been tested properly in terms of activity measurements, strength testing or migration of implants. There is diversity in the literature regarding whether tibial component with too much deviation from a neutral axis can lead to increased migration and eventually aseptic solution. To date, only a few trials, with diverging results, have assessed migration of the implants implanted with KA or FA. The methods are so far perceived as controversial, despite the widespread use.

KA or FA can be performed by manual conventional surgery; however, the newly introduced robotic assisted surgery probably yields higher accuracy and precision of the cuts during surgery. This makes robotic assisted surgery well suited for personalized surgery. Yet, it is claimed that because of diversity of the different features for planning and executing the surgery, each system should be evaluated separately, and not as a group. The investigators therefore planned this study to assess the efficacy of robotic assisted surgery comparing MA and personalized alignment (PA) techniques.

Aims of the trial

1. Evaluate the clinical outcomes of patients who have had TKA with PA and compare it with conventional MA.
2. Analyse and compare the in vivo stability over time of TKA operated with PA vs. MA using CT- based radiostereometric analysis (CT-RSA).
3. Evaluate the postoperative position of the implants using two different alignment philosophies.

Objective Perform TKAs on patients using ROSA® Knee System (Zimmer Biomet, Warsaw, Indiana USA) robotic assisted surgery and randomize the patients to either PA or MA.

Materials and methods

A multiple blinded randomized controlled parallel superiority trial will be performed, where the patients, study nurse, statistician and physiotherapists are blinded to the surgical method (PA or MA). The study will include 152 patients. The study adheres to the consort statement.

Surgery All surgeons involved in the trial are experienced knee surgeons. The surgeons have received thorough tutoring in the use of the ROSA Knee System and the Persona TKA, and both alignment techniques have now been adopted in our standard treatment of end stage OA. The learning curve of robotic assisted surgery is probably very small, and more related to time spent on the procedure rather than placement of the implants. The placement of the tibial implant will be restricted in the coronal plane to maximum 5 degrees of varus and 2 degrees of valgus. In sagittal plane, the slope will be limited to between 0-10 degrees.

The Persona TKA implant although contemporary, is a well-documented implant with very low migration.

The MA and PA techniques are well known and already used in a widespread fashion all around the world. Several clinics in Norway have also adopted the methods.

Implantation of tantalum markers in bone and polyethylene has been performed for more than 40 years in numerous studies without any known complications.

Known but rare complications to robotic surgery are fractures at the site of insertion of the bone pins, and pin site infections. In elderly or osteoporotic patients, the surgeons will consider using unicortical engagement of the pins. Concerning infections, all the default precautions in the OR will be taken, such as preoperative and postoperative administration of antibiotics, strict sterile procedures etc.

ELIGIBILITY:
Inclusion Criteria:

• femoro-tibial or patello-femoral osteoarthritis (Kellgren-Lawrence, K-L) grade 2-4 with persistent pain, referred to Kristiansund Hospital for primary TKA

Exclusion Criteria:

* serious psychiatric disorders
* dementia
* drug abuse
* patients not able to speak and read Norwegian language making them noncompliant or unable to perform an informed consent
* Patients with ongoing cancer therapy
* Patients with ASA (The American Society of Anesthesiologists physical status class risk stratification system) classification >3
* Patients in the need of walking aid devices
* Patients in need of primary revision arthroplasty or more than 15 degrees of varus or 5 degrees of valgus on preoperative HKA images.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2035-05-01 (Estimated)

PRIMARY OUTCOMES:
MTPM | 2 years
  Maximum Total Point Motion measured by CT -based RSA in millimeters.

SECONDARY OUTCOMES:
XYZ translation | 2 years
  Translation of implant measured by CT -based RSA in millimeters
XYZ rotation | 2 years
  Rotation of implant measured by CT -based RSA in degrees
Steps per day | 1 year and 2 years
  ActivePAL accelerator registration of mean steps per day measured 24/7 for a week
Walking speed | 1 and 2 years
  ActivePAL accelerator registration of mean meter per second measured 24/7 for a week
Stair climbing | 1 and 2 years
  Standardized climbing and descending of stairs up and down. Time in seconds measured up, down and total.
Maximal voluntary contraction flexion | 1 and 2 years
  Isometric contraction at 90 degrees knee flexion measured in Newtons with Tindeq force cell
Maximal voluntary contraction extension | 1 and 2 years
  Isometric contraction at 90 degrees knee extension measured in Newtons with Tindeq force cell
Maximal voluntary contraction | 1 and 2 years
  Isometric contraction at 90 degrees knee flexion measured in Newtons with Tindeq force cell
Sit to stand test | 1 and 2 years
  Maximum number of repetitive transitions from sitting on a chair to standing without the use of hands during 30 seconds
KOOS score | 1 and 2 years
  Knee Injury and Osteoarthritis of 5 dimensions measuring activity of daily living (ADL), Quality of life, Sport and recreation, pain and symptoms. From 0 (bad) to 100 (excellent)
FJS | 1 and 2 years
  Forgotten Joint Score is a 12 item scale assessing the ability to forget the operated joint as artificial during activities of daily living. Ranges from 0 (bad) to 100 (excellent)
Eq-5D | 1 and 2 years
  EuroQol 5 Dimensions is a generic patient reported outcome measure measuring quality of life. The scale ranges from 100 ('the best imaginable health state') to 0 ('the worst imaginable health state' ).
VAS | 1 and 2 years
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')

CONTACTS AND LOCATIONS:
Overall Officials: Frank-David Øhrn, MD, PhD, Study Director — Møre og Romsdal Hospital Trust; Kirsti Sevaldsen, MD, PhD, Study Chair — Møre og Romsdal Hospital Trust
Locations (1):
- Kristiansund Hospital, Møre and Romsdal Hospital Trust, Kristiansund, Møre and Romsdal, Norway

IPD SHARING:
Plan to Share IPD: Yes
Upon proper request to the corresponding author data will be shared anonymously.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and for 2 years

REFERENCES:
- [Background] Bellemans J, Colyn W, Vandenneucker H, Victor J. The Chitranjan Ranawat award: is neutral mechanical alignment normal for all patients? The concept of constitutional varus. Clin Orthop Relat Res. 2012 Jan;470(1):45-53. doi: 10.1007/s11999-011-1936-5. PMID 21656315
- [Background] Lee YS, Howell SM, Won YY, Lee OS, Lee SH, Vahedi H, Teo SH. Kinematic alignment is a possible alternative to mechanical alignment in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3467-3479. doi: 10.1007/s00167-017-4558-y. Epub 2017 Apr 24. PMID 28439636
- [Background] Begum FA, Kayani B, Magan AA, Chang JS, Haddad FS. Current concepts in total knee arthroplasty : mechanical, kinematic, anatomical, and functional alignment. Bone Jt Open. 2021 Jun;2(6):397-404. doi: 10.1302/2633-1462.26.BJO-2020-0162.R1. PMID 34139884
- [Background] Lustig S, Sappey-Marinier E, Fary C, Servien E, Parratte S, Batailler C. Personalized alignment in total knee arthroplasty: current concepts. SICOT J. 2021;7:19. doi: 10.1051/sicotj/2021021. Epub 2021 Mar 26. PMID 33812467
- [Background] Liu B, Feng C, Tu C. Kinematic alignment versus mechanical alignment in primary total knee arthroplasty: an updated meta-analysis of randomized controlled trials. J Orthop Surg Res. 2022 Apr 4;17(1):201. doi: 10.1186/s13018-022-03097-2. PMID 35379289
- [Background] Hasan S, Kaptein BL, Nelissen RGHH, van Hamersveld KT, Toksvig-Larsen S, Marang-van de Mheen PJ. The Influence of Postoperative Coronal Alignment on Tibial Migration After Total Knee Arthroplasty in Preoperative Varus and Valgus Knees: A Secondary Analysis of 10 Randomized Controlled Trials Using Radiostereometric Analysis. J Bone Joint Surg Am. 2021 Dec 15;103(24):2281-2290. doi: 10.2106/JBJS.20.01659. PMID 34648477
- [Background] van Hamersveld KT, Marang-van de Mheen PJ, Nelissen RGHH. The Effect of Coronal Alignment on Tibial Component Migration Following Total Knee Arthroplasty: A Cohort Study with Long-Term Radiostereometric Analysis Results. J Bone Joint Surg Am. 2019 Jul 3;101(13):1203-1212. doi: 10.2106/JBJS.18.00691. PMID 31274722
- [Background] Laende EK, Richardson CG, Dunbar MJ. A randomized controlled trial of tibial component migration with kinematic alignment using patient-specific instrumentation versus mechanical alignment using computer-assisted surgery in total knee arthroplasty. Bone Joint J. 2019 Aug;101-B(8):929-940. doi: 10.1302/0301-620X.101B8.BJJ-2018-0755.R3. PMID 31362561
- [Background] Choi BS, Kim SE, Yang M, Ro DH, Han HS. Functional alignment with robotic-arm assisted total knee arthroplasty demonstrated better patient-reported outcomes than mechanical alignment with manual total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):1072-1080. doi: 10.1007/s00167-022-07227-5. Epub 2022 Nov 15. PMID 36378291
- [Background] Vermue H, Batailler C, Monk P, Haddad F, Luyckx T, Lustig S. The evolution of robotic systems for total knee arthroplasty, each system must be assessed for its own value: a systematic review of clinical evidence and meta-analysis. Arch Orthop Trauma Surg. 2023 Jun;143(6):3369-3381. doi: 10.1007/s00402-022-04632-w. Epub 2022 Sep 25. PMID 36153769
- [Background] Petersen ET, Rytter S, Koppens D, Dalsgaard J, Hansen TB, Andersen MS, Stilling M. Medial congruent polyethylene design show different tibiofemoral kinematics and enhanced congruency compared to a standard symmetrical cruciate retaining design for total knee arthroplasty-an in vivo randomized controlled study of gait using dynamic radiostereometry. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):933-945. doi: 10.1007/s00167-022-07036-w. Epub 2022 Jul 9. PMID 35809105
- [Background] Scott G, Imam MA, Eifert A, Freeman MA, Pinskerova V, Field RE, Skinner J, Banks SA. Can a total knee arthroplasty be both rotationally unconstrained and anteroposteriorly stabilised? A pulsed fluoroscopic investigation. Bone Joint Res. 2016 Mar;5(3):80-6. doi: 10.1302/2046-3758.53.2000621. PMID 26965166
- [Background] Mathijssen NMC, Verburg H, London NJ, Landsiedl M, Dominkus M. Patient reported outcomes and implant survivorship after Total knee arthroplasty with the persona knee implant system: two year follow up. BMC Musculoskelet Disord. 2019 Mar 4;20(1):97. doi: 10.1186/s12891-019-2470-y. PMID 30832636
- [Background] Christensson A, Tveit M, Kesteris U, Flivik G. Similar migration for medial congruent and cruciate-retaining tibial components in an anatomic TKA system: a randomized controlled trial of 60 patients followed with RSA for 2 years. Acta Orthop. 2022 Jan 3;93:68-74. doi: 10.1080/17453674.2021.1983709. PMID 34633885
- [Background] Koster LA, Meinardi JE, Kaptein BL, Van der Linden-Van der Zwaag E, Nelissen RGHH. Two-year RSA migration results of symmetrical and asymmetrical tibial components in total knee arthroplasty: a randomized controlled trial. Bone Joint J. 2021 May;103-B(5):855-863. doi: 10.1302/0301-620X.103B5.BJJ-2020-1575.R2. PMID 33934647
- [Background] Tuecking LR, Savov P, Zander M, Jeremic D, Windhagen H, Ettinger M. Comparable accuracy of femoral joint line reconstruction in different kinematic and functional alignment techniques. Knee Surg Sports Traumatol Arthrosc. 2023 Sep;31(9):3871-3879. doi: 10.1007/s00167-023-07360-9. Epub 2023 Mar 14. PMID 36917247
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Kersten P, Kucukdeveci AA, Tennant A. The use of the Visual Analogue Scale (VAS) in rehabilitation outcomes. J Rehabil Med. 2012 Jun;44(7):609-10. doi: 10.2340/16501977-0999. No abstract available. PMID 22674245
- [Background] Shim J, Hamilton DF. Comparative responsiveness of the PROMIS-10 Global Health and EQ-5D questionnaires in patients undergoing total knee arthroplasty. Bone Joint J. 2019 Jul;101-B(7):832-837. doi: 10.1302/0301-620X.101B7.BJJ-2018-1543.R1. PMID 31256677
- [Background] Allen GM, Gandevia SC, McKenzie DK. Reliability of measurements of muscle strength and voluntary activation using twitch interpolation. Muscle Nerve. 1995 Jun;18(6):593-600. doi: 10.1002/mus.880180605. PMID 7753121
- [Background] Unhjem R, van den Hoven LT, Nygard M, Hoff J, Wang E. Functional Performance With Age: The Role of Long-Term Strength Training. J Geriatr Phys Ther. 2019 Jul/Sep;42(3):115-122. doi: 10.1519/JPT.0000000000000141. PMID 28786909
- [Background] Petersson N, Langgard Jorgensen S, Kjeldsen T, Mechlenburg I, Aagaard P. Blood Flow Restricted Walking in Elderly Individuals with Knee Osteoarthritis: A Feasibility Study. J Rehabil Med. 2022 Jun 20;54:jrm00282. doi: 10.2340/jrm.v54.2163. PMID 35266006
- [Background] Engseth LHW, Schulz A, Pripp AH, Rohrl SMH, Ohrn FD. CT-based migration analysis is more precise than radiostereometric analysis for tibial implants: a phantom study on a porcine cadaver. Acta Orthop. 2023 Apr 27;94:207-214. doi: 10.2340/17453674.2023.12306. PMID 37114404
- [Background] Ohrn FD, Lian OB, Tsukanaka M, Rohrl SM. Early migration of a medially stabilized total knee arthroplasty : a radiostereometric analysis study up to two years. Bone Jt Open. 2021 Sep;2(9):737-744. doi: 10.1302/2633-1462.29.BJO-2021-0115.R1. PMID 34493056
- [Background] Garling EH, Kaptein BL, Geleijns K, Nelissen RG, Valstar ER. Marker Configuration Model-Based Roentgen Fluoroscopic Analysis. J Biomech. 2005 Apr;38(4):893-901. doi: 10.1016/j.jbiomech.2004.04.026. PMID 15713311
- [Background] Laur O, Weaver MJ, Bridge C, Chow E, Rosenthal M, Bay C, Javedan H, Harris MB, Khurana B. Computed tomography-based body composition profile as a screening tool for geriatric frailty detection. Skeletal Radiol. 2022 Jul;51(7):1371-1380. doi: 10.1007/s00256-021-03951-0. Epub 2021 Dec 4. PMID 34862921
- [Background] Van Leeuwen JAMJ, Snorrason F, Rohrl SM. No radiological and clinical advantages with patient-specific positioning guides in total knee replacement. Acta Orthop. 2018 Feb;89(1):89-94. doi: 10.1080/17453674.2017.1393732. Epub 2017 Nov 22. PMID 29161930
- [Background] Husby VS, Rian T, Klaksvik J, Wik TS, Winther SB. Physical activity in the first postoperative week in 132 knee arthroplasty patients randomized to 3 different analgesic regimens. Medicine (Baltimore). 2023 Apr 21;102(16):e33471. doi: 10.1097/MD.0000000000033471. PMID 37083790
- [Background] Bin Sheeha B, Granat M, Williams A, Johnson DS, Jones R. Does free-living physical activity improve one-year following total knee arthroplasty in patients with osteoarthritis: A prospective study. Osteoarthr Cartil Open. 2020 Apr 13;2(3):100065. doi: 10.1016/j.ocarto.2020.100065. eCollection 2020 Sep. PMID 36474675
- [Background] Husby VS, Helgerud J, Bjorgen S, Husby OS, Benum P, Hoff J. Early maximal strength training is an efficient treatment for patients operated with total hip arthroplasty. Arch Phys Med Rehabil. 2009 Oct;90(10):1658-67. doi: 10.1016/j.apmr.2009.04.018. PMID 19801053
- [Background] Pijls BG, Valstar ER, Nouta KA, Plevier JW, Fiocco M, Middeldorp S, Nelissen RG. Early migration of tibial components is associated with late revision: a systematic review and meta-analysis of 21,000 knee arthroplasties. Acta Orthop. 2012 Dec;83(6):614-24. doi: 10.3109/17453674.2012.747052. Epub 2012 Nov 9. PMID 23140091
- [Background] Derbyshire B, Prescott RJ, Porter ML. Notes on the use and interpretation of radiostereometric analysis. Acta Orthop. 2009 Feb;80(1):124-30. doi: 10.1080/17453670902807474. PMID 19234894
- [Background] Masse V, Cholewa J, Shahin M. Personalized alignment for total knee arthroplasty using the ROSA(R) Knee and Persona(R) knee systems: Surgical technique. Front Surg. 2023 Jan 10;9:1098504. doi: 10.3389/fsurg.2022.1098504. eCollection 2022. PMID 36733674
- [Background] Clement ND, Al-Zibari M, Afzal I, Deehan DJ, Kader D. A systematic review of imageless hand-held robotic-assisted knee arthroplasty: learning curve, accuracy, functional outcome and survivorship. EFORT Open Rev. 2020 May 9;5(5):319-326. doi: 10.1302/2058-5241.5.190065. eCollection 2020 May. PMID 32509337
- [Background] Schopper C, Proier P, Luger M, Gotterbarm T, Klasan A. The learning curve in robotic assisted knee arthroplasty is flattened by the presence of a surgeon experienced with robotic assisted surgery. Knee Surg Sports Traumatol Arthrosc. 2023 Mar;31(3):760-767. doi: 10.1007/s00167-022-07048-6. Epub 2022 Jul 21. PMID 35864240
- [Background] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Ohrn FD, Engseth LHW, Pripp AH, Rohrl SMH, Schulz A. Dose reduction does not impact the precision of CT-based RSA in tibial implants: a diagnostic accuracy study on precision in a porcine cadaver. Acta Orthop. 2023 Oct 31;94:550-544. doi: 10.2340/17453674.2023.24022. PMID 37909103
- See also: Consort Statement — http://view.officeapps.live.com/op/view.aspx?src=https%3A%2F%2Fwww.equator-network.org%2Fwp-content%2Fuploads%2F2017%2F05%2FCONSORT-2010-Checklist.doc&wdOrigin=BROWSELINK
- See also: ASA classification system — http://www.asahq.org/standards-and-practice-parameters/statement-on-asa-physical-status-classification-system

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT06507046/Prot_SAP_000.pdf